CLINICAL TRIAL: NCT06880367
Title: Neuromodulatory Effects of Audio-proprio-phonatory Reinforcement Training on Subjective Tinnitus, Demonstrated by High-density Electroencephalogram (HD EEG)
Acronym: PHONACOU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: CHUO-2024-18
Record Dates: First submitted 2025-03-06; First posted 2025-03-17 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Tinnitus, Subjective
Keywords: Subjective tinnitus; neuromodulation; audio-proprio-phonatory reinforcement; high-density electroencephalogram
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Intervention Model Description: This study is prospective, randomized into two groups with stratification based on the THI score specifically comparing grade 3 to grades 4 and 5.
  The neurology staff conducting the HD EEG examination will remain unaware of the treatment allocation, ensuring a single-blinded design.
Who Masked: Care Provider
Masking Description: Neurology staff performing the HD EEG examination will not know the treatment arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: audio-proprio-phonatory training (phase 1) then no training (phase 2) (Experimental): Patients will undergo audio-proprio-phonatory training and evaluate their discomfort using the VAS-D scale for a duration of five weeks. Following this period, they will be assessed with the THI score and undergo HD EEG examination (T1). Subsequently, there will be no training and patients will again evaluate their discomfort using the VAS-D score over the next five weeks. At the conclusion of the ten weeks of follow-up, patients will be assessed with the THI score.
  Interventions: Behavioral: The intervention is an audio-proprio-phonatory training; Diagnostic Test: high-density electroencephalogram (HD-EEG)
- Group 2: No training (phase 1) then audio-proprio-phonatory training (phase 2) (Experimental): Patients will be no training and evaluate their discomfort using the VAS-D scale for a duration of five weeks. Following this period, they will be assessed with the THI score and undergo HD EEG examination (T1). Subsequently, there will undergo audio-proprio-phonatory training and patients will again evaluate their discomfort using the VAS-D score over the next five weeks. At the conclusion of the ten weeks of follow-up, patients will be assessed with the THI score.
  Interventions: Behavioral: The intervention is an audio-proprio-phonatory training; Diagnostic Test: high-density electroencephalogram (HD-EEG)

INTERVENTIONS:
Behavioral: The intervention is an audio-proprio-phonatory training — The audio-proprio-phonatory training involves engaging in group workshops and performing exercise sessions independently, following the guidance provided by the specialist, over a duration of five weeks
Diagnostic Test: high-density electroencephalogram (HD-EEG) — HD-EEG examination with 256 channels distributed throughout the skull that record resting brain connectivity(10 min).

SUMMARY:
Our ecological approach to neuromodulation in the field of "acouphonology" empowers tinnitus patients to act as their own source of sound stimuli through audio-proprio-phonatory reinforcement (APPR). By engaging in self-phonations, individuals uncoverthe vast potential for sound production, which can effectively mask their tinnitus or induce residual inhibition, all without relying on external sources.

This clinical study aims to illustrate the positive impact of audio-proprio-phonatory reinforcement training on individuals suffering from chronic subjective tinnitus. This will be further supported and quantified through high-definition electroencephalography (HD EEG) as we explore the relationship between changes in connectivity within specific brain regions and the varying degrees of response to the therapeutic protocol.

DETAILED DESCRIPTION:
Three visits will be conducted, with intervals of two periods lasting five weeks each.

Inclusion visit (T0): Following the assessment of eligibility, the patient will receive an informative document regarding the study. After a period of contemplation, the patient will provide consent to participate.

This visit will include a medical examination, an APPR test accompagnied by spectrogram feedback, a tinnitus assessment focusing on residual inhibition, high-density electroencephalograms and self-assessment questionnaires.

Phase 1: Other the course of five weeks, Group A, designated for"audio-proprio-phonatory training" will participate in one group videoconference session each week, along with daily exercises to complete. Participants will also be required to self-assess using the Visual Analog Scale of discomfort (VAS-D) on the days of the group workshops and on Fridays (both morning and evening).

Concurrently, Group B, labeled "no training" will conduct self-assessments using the VAS-D on Mondays and Fridays (morning and evening).

T1 visit: This visit will involve a medical examination, high-density electroencephalograms and self-assessment questionnaires will be performed.

Phase 2: The 2 groups will switch roles and follow the same protocol as outlined in phase 1.

End of study visit (T2): A medical examination and self-assessment questionnaires will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Person who agreed to participate in the study and gave consent
* Aged ≥ 18 years and < 85 years
* Suffering from subjective tinnitus for more than 3 months
* Have a score on the THI questionnaire taken at T0 greater than or equal to 38
* Be equipped with a smartphone compatible with the Siopi application and a computer connection for videoconference sessions
* Have answered the questionnaires on the Siopi application: THI, VAS-D and associated questions and insomnia severity index
* Have committed to diligently following the study protocol, including independent training
* Have agreed not to take other new treatments for tinnitus throughout the duration of the study
* Able to understand and carry out assessment instructions.

Exclusion Criteria:

* Patient suffering from objective tinnitus
* Current port of white noise generators
* Patient having consulted phoniatrics more than twice or having participated in more than two sound-mediated workshop sessions
* Bilateral hearing loss > 40 dB uncorrected on an audiogram or having declared serious or severe hearing loss on Siopi questionnaire, with or without prosthetic correction
* New therapy introduced less than 2 months ago
* Psychatric disorders causing auditory hallucinations
* Protected person (under guardianship or curatorship)
* Person under judicial protection
* Person deprived of liberty
* Person not affiliated to a social security system
* Pregnant or breastfeeding woman
* Person participating in a drug study

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2028-09-18 (Estimated); Study Completion 2028-09-18 (Estimated)

PRIMARY OUTCOMES:
The objective is to assess whether training that incorporates audio-proprio-phonatory reinforcement (APPR) can alleviate the daily life disability associated with tinnitus, in comparison to patients who have not undergo APPR training. | Evaluation at T0 (Day 0) and T1 (Day 42 +/- 7 days) of the study.
  The international Tinnitus Handicap Inventory (THI) questionnaire will be employed to assess the influence of training on the quality of patients affected by tinnitus.. This assessment will include a comparison of the changes in THI scores from T0 (Day 0) to T1 (Day 42) in the group that underwent APPR training, relative to the changes in THI scores from T0 (Day 0) to T1 (Day 42) in the group that did not receive APPR training.

SECONDARY OUTCOMES:
Determine whether APPR exercises reduce the discomfort linked to tinnitus in the short term (tinnitus discomfort VAS), compared to patients who have not followed APPR training | Evaluation at T0 (Day 0), T1 (Day 42 +/- 7 days) and T2 (Day 92 +/- 7 days)
  Visual analog scale of discomfort (VAS-D) tinnitus (scale from 0 to 10 with 10 being the worst score), completed by the patient (on the Siopi application), weekly between T0 (Day 0) and T1 (Day 42), 4 times per week.
  * For the group with APPR training between T0 and T1, they will be completed : morning and evening, on the day of the group workshops (Monday or Tuesday) and on Friday
  * For the group without APPR training between T0 et T1, they will be completed : upon waking up and in the evening, every Monday and Friday.
  This will first involve comparing the average of the daily differences obtained over 5 weeks . Then we will compare the evolution (taking the daily average of the tinnitus VAS-D) over 5 weeks between T0 et T1 for the 2 groups.
  NB : These results can be confirmed bu analyzing the tinnitus VAS-D over the 5 weeks between T1 (Day 42) and T2 (Day 92) for group B (having the APPR training over this period.
Study the stability over time of quality of life (THI score) after APPR training. | Evaluation at T1 (Day 42 +/- 7 days) and T2 (Day 92 +/- 7 days)
  To study stability over time, only data from patients in group A, without APPR training between T1 (Day 42) et T2 (Day 92) will be used :
  - The THI score (scale from 0 to 100 with 10 being the worst score) measured at T1 and T2 This will involve comparing the results at T2 compared to T1.
Study the stability over time of tinnitus-related discomfort (VAS) after APPR training. | Evaluation at T1 (Day 42 +/- 7 days) and T2 (Day 92 +/- 7 days)
  To study stability over time, only data from patients in group A, without APPR training between T1 (Day 42) et T2 (Day 92) will be used :
  - VAS-D tinnitus scale (scale from 0 to 10 with 10 being the worst score), completed by te patient (on the Siopi application), weekly between T1 and T2, 4 times per week.
Describe the evolution of quality of life (THI score) during the study | Evaluation at T0 (Day 0), T1 (Day 42 +/- 7 days) and T2 (Day 92 +/- 7 days)
  Evolution over time of the THI score (scale from 0 to 100 with 10 being the worst score) measured at T0 (Day 0), T1 (Day 42) and T2 (Day 92) for the 2 groups.
Describe the evolution of other collateral discomfort (noise) to tinnitus of patients who followed APPR training, compared to patients without APPR training | Evaluation at T0 (Day 0), T1 (Day 42 +/- 7 days) and T2 (Day 92 +/- 7 days)
  Visual analog scale VAS-D (scale from 0 to 10 with 10 being the worst score) associated questions about noises, completed by the patient (on the Siopi application), weekly between T0 (Day 0) and T1 (Day 42), at a rate of 4 times per week, for the 2 groups. We will compare the evolution of each VAS-D taken independantly, taking the daily average of VAS-D concerned, over the 5 weeks between T0 and T1 for the 2 groups.
Describe the evolution of other collateral discomfort (cervical pain) to tinnitus of patients who followed APPR training, compared to patients without APPR training | Evaluation at T0 (Day 0), T1 (Day 42 +/- 7 days) and T2 (Day 92 +/- 7 days)
  Visual analog scale VAS-D (scale from 0 to 10 with 10 being the worst score) associated questions with cervical pain completed by the patient (on the Siopi application), weekly between T0 (Day 0) and T1 (Day 42), at a rate of 4 times per week, for the 2 groups. We will compare the evolution of each VAS-D taken independantly, taking the daily average of VAS-D concerned, over the 5 weeks between T0 and T1 for the 2 groups.
Describe the evolution of other collateral discomfort (jaw pain) to tinnitus of patients who followed APPR training, compared to patients without APPR training | Evaluation at T0 (Day 0), T1 (Day 42 +/- 7 days) and T2 (Day 92 +/- 7 days)
  Visual analog scale VAS-D (scale from 0 to 10 with 10 being the worst score) associated questions with jaw pain completed by the patient (on the Siopi application), weekly between T0 (Day 0) and T1 (Day 42), at a rate of 4 times per week, for the 2 groups. We will compare the evolution of each VAS-D taken independantly, taking the daily average of VAS-D concerned, over the 5 weeks between T0 and T1 for the 2 groups.
Describe the evolution of other collateral discomfort (sleep) to tinnitus of patients who followed APPR training, compared to patients without APPR training | Evaluation at T0 (Day 0), T1 (Day 42 +/- 7 days) and T2 (Day 92 +/- 7 days)
  Visual analog scale VAS-D (scale from 0 to 10 with 10 being the worst score) associated questions about sleep completed by the patient (on the Siopi application), weekly between T0 (Day 0) and T1 (Day 42), at a rate of 4 times per week, for the 2 groups. We will compare the evolution of each VAS-D taken independantly, taking the daily average of VAS-D concerned, over the 5 weeks between T0 and T1 for the 2 groups.
Describe the evolution of other collateral discomfort(stress-anxiety) to tinnitus of patients who followed APPR training, compared to patients without APPR training | Evaluation at T0 (Day 0), T1 (Day 42 +/- 7 days) and T2 (Day 92 +/- 7 days)
  Visual analog scales VAS-D (scale from 0 to 10 with 10 being the worst score) associated questions about stress-anxiety completed by the patient (on the Siopi application), weekly between T0 (Day 0) and T1 (Day 42), at a rate of 4 times per week, for the 2 groups. We will compare the evolution of each VAS-D taken independantly, taking the daily average of VAS-D concerned, over the 5 weeks between T0 and T1 for the 2 groups.
Evaluate the effect of APPR training on the usual connectivity of HD-EEG, compared to patients who did not follow APPR training | Evaluation at T0 (Day 0) and T1 (Day 42 +/- 7 days)
  Exploratory analyzes of the different HD-EEG parameters measured at T0 (Day 0) and T1 (Day 42) in the 2 groups :
  The evolution of HD-EEG connectivity such as : network efficiency, dwill be described in the group with APPR training and compared to the evolution of this same parameter in the group without APPR training between T0 and T1.
Evaluate the effect of APPR training on the usual connectivity (duration of states) of HD-EEG, compared to patients who did not follow APPR training | Evaluation at T0 (Day 0) and T1 (Day 42 +/- 7 days)
  Exploratory analyzes of the different HD-EEG parameters measured at T0 (Day 0) and T1 (Day 42) in the 2 groups :
  The evolution of HD-EEG microstate parameters such as : duration of states, will be described in the group with APPR training and compared to the evolution of this same parameter in the group without APPR training between T0 and T1.
Evaluate the effect of APPR training on the usual microstate parameters (distribution of states) of HD-EEG, compared to patients who did not follow APPR training | Evaluation at T0 (Day 0) and T1 (Day 42 +/- 7 days)
  Exploratory analyzes of the different HD-EEG parameters measured at T0 (Day 0) and T1 (Day 42) in the 2 groups :
  The evolution of HD-EEG connectivity and microstate parameters such as : distribution of states, will be described in the group with APPR training and compared to the evolution of this same parameter in the group without APPR training between T0 and T1.
Describe the evolution of the quality of life (THI score) of patients before and after APPR training and the usual connectivity and microstate parameters of HD-EEG, over time. | Evaluation at T0 (Day 0) and T1 (Day 42 +/- 7 days)
  Exploratory analyzes of the search for correlation between evolution of connectivity parameters of HD-EEG (determine specific parameters like distribution of states) with the evolution of THI score (scale from 0 to 100 with 100 being the worst score) will be explored (between T0 and T1)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Dr MARIE-BAILLY, PhD, Principal Investigator — CHU Orléans
Locations (1):
- CHU Orleans, Orléans, France

REFERENCES:
- [Background] Norena AJ. An integrative model of tinnitus based on a central gain controlling neural sensitivity. Neurosci Biobehav Rev. 2011 Apr;35(5):1089-109. doi: 10.1016/j.neubiorev.2010.11.003. Epub 2010 Nov 19. PMID 21094182
- [Background] Tonndorf J. The analogy between tinnitus and pain: a suggestion for a physiological basis of chronic tinnitus. Hear Res. 1987;28(2-3):271-5. doi: 10.1016/0378-5955(87)90054-2. PMID 2820913
- [Background] De Ridder D, Vanneste S, Weisz N, Londero A, Schlee W, Elgoyhen AB, Langguth B. An integrative model of auditory phantom perception: tinnitus as a unified percept of interacting separable subnetworks. Neurosci Biobehav Rev. 2014 Jul;44:16-32. doi: 10.1016/j.neubiorev.2013.03.021. Epub 2013 Apr 15. PMID 23597755
- [Background] Huang H, Cai Y, Feng X, Li Y. [An electroencephalogram-based study of resting-state spectrogram and attention in tinnitus patients]. Sheng Wu Yi Xue Gong Cheng Xue Za Zhi. 2021 Jun 25;38(3):492-497. doi: 10.7507/1001-5515.202012015. Chinese. PMID 34180194
- [Background] Vanneste S, Byczynski G, Verplancke T, Ost J, Song JJ, De Ridder D. Switching tinnitus on or off: An initial investigation into the role of the pregenual and rostral to dorsal anterior cingulate cortices. Neuroimage. 2024 Aug 15;297:120713. doi: 10.1016/j.neuroimage.2024.120713. Epub 2024 Jun 27. PMID 38944171